CLINICAL TRIAL: NCT03931902
Title: The Comparison of Laryngeal Mask Airway and Endotracheal Tube in Premature Neonates Undergoing General Anesthesia for Inguinal Hernia Repair Surgery
Brief Title: The Comparison of Laryngeal Mask Airway and Endotracheal Tube in General Anesthesia for Premature Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20190017
Record Dates: First submitted 2019-04-23; First posted 2019-04-30 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2020-12

CONDITIONS: Preterm Infant; Anesthesia; Respiratory Complication
Keywords: pediatric airway management
MeSH Terms: conditions — Premature Birth | interventions — Intubation; Laryngeal Masks

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laryngeal Mask Airway (LMA) (Experimental): Using laryngeal mask airway as the airway device during general anesthesia
  Interventions: Device: intubation with laryngeal mask airway
- Endotracheal Tube (ETT) (Active Comparator): Using endotracheal tube as the airway device during general anesthesia
  Interventions: Device: intubation with Endotracheal tube

INTERVENTIONS:
Device: intubation with Endotracheal tube — After masking ventilation with sevoflurane till the adequate anesthetic depth, intubation will be done with endotracheal tube (ETT).
  Arms: Endotracheal Tube (ETT)
Device: intubation with laryngeal mask airway — After masking ventilation with sevoflurane till the adequate anesthetic depth, intubation will be done with laryngeal mask airway (LMA).
  Arms: Laryngeal Mask Airway (LMA)

SUMMARY:
Objectives: To compare the perioperative respiratory adverse events between using laryngeal mask airway and endotracheal tube in preterm neonates receiving general anesthesia for hernia surgery.

DETAILED DESCRIPTION:
The participant patients will be randomly allocated into two groups: the laryngeal mask airway group (LMA group) and endotracheal tube group (ETT group). Masking ventilation with sevoflurane will be used for anesthesia induction till the adequate anesthetic depth. Intubation with laryngeal mask airway (LMA) or endotracheal tube (ETT) will be done as allocated group. After the surgery completed and the patient wakened up, the anesthesiologist will remove the LMA or ETT according to the clinical criteria for extubation.

ELIGIBILITY:
Inclusion Criteria:

* preterm neonates (gestational age < 37 weeks) in our neonatal ward scheduled to receive unilateral or bilateral inguinal hernia repair surgery, and whose body weight > 2000g at surgery

Exclusion Criteria:

* emergent surgery, infants who was intubated before surgery, long-term oxygen or mechanical ventilation dependence, severe congenital cardiopulmonary disease, lacking of birth history, combination with other major surgery, postmenstrual age > 52 weeks at surgery

Max Age: 52 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Perioperative respiratory complication | from induction of anesthesia to postoperative 24 hours
  laryngospasm, bronchospasm, severe cough, delayed extubation or prolonged oxygen dependence, apnea, bradycardia, and postoperative stridor
postoperative hospital stays | from postoperative day 1 up to postoperative day 30
  the lengths of postoperative hospital stays

CONTACTS AND LOCATIONS:
Overall Officials: Miaopei Su, Master, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No